CLINICAL TRIAL: NCT00223236
Title: A Double-blind, Placebo-controlled Trial of Citicoline add-on Therapy in Patients With a History of Mania or Hypomania and Cocaine Abuse/Dependence
Brief Title: Trial of Citicoline Therapy in Patients With Mania or Hypomania and Cocaine Abuse/Dependence
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Sherwood Brown, professor, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 03T-439
Record Dates: First submitted 2005-09-15; First posted 2005-09-22 (Estimated); Results first posted 2014-08-11 (Estimated); Last update posted 2014-08-11 (Estimated); Status verified 2014-08

CONDITIONS: Mania; Hypomania; Cocaine Abuse; Cocaine Dependence
MeSH Terms: conditions — Mania; Cocaine-Related Disorders | interventions — Cytidine Diphosphate Choline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Citicoline (Active Comparator): Citicoline is an over the counter supplement that may have neuroprotective properties and may have antidepressant effects.
  Interventions: Drug: Citicoline
- Placebo (Placebo Comparator): Inactive ingredient matching the active medication in appearance
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Citicoline — Citicoline or placebo will be given beginning at one table (500mg)/day with an increase to two tablets (1000mg)/day at week 2, three tablets (1500mg)/day at week 4 and four tablets (2000mg)/day at week 6. Patients will remain on 2000mg/day through week 12. Doses will be decreased if needed due to side effects.
  Other Names: Cytidine-5'-diphosphocholine; CDP-choline
  Arms: Citicoline
Drug: Placebo — Placebo matching active medication in all other aspects.
  Other Names: Identical placebo
  Arms: Placebo

SUMMARY:
The purpose of this research is to determine if a citicoline supplement is associated with a reduction in cocaine use and craving in patients with bipolar disorder (a mental disorder marked by alternating periods of mania and depression) or schizoaffective disorder/bipolar type (a psychotic disturbance in which there is a mixture of schizophrenic and manic-depressive symptoms) and cocaine abuse/dependence. This research also wants to explore if citicoline supplements are associated with greater improvement in symptoms of mania and on memory and cognition (the mental faculty of perception, reasoning, and judgement) in these patients.

DETAILED DESCRIPTION:
Forty-four outpatients meeting the inclusion and exclusion criteria were enrolled after completing an Institutional Review Board (IRB)-approved informed consent process. Baseline evaluation included a medical and psychiatric history, structured diagnostic interview using Diagnostic and Statistical Manual (DSM)-IV criteria, mood assessment with the Inventory of Depressive Symptomatology-Self Report (IDS-SR), Young Mania Rating Scale (YMRS), and cognitive assessment with the Rey Auditory Verbal Learning Test (RAVLT). Alternate but equivalent versions of the RAVLT were used to minimize practice effects with repeated administration. Cocaine use was assessed at each biweekly visit with urine drug screens. Citicoline or placebo was given beginning at one tablet (500 mg)/day with an increase to two tablets (1000 mg/day) at week 2, three tablets (1500 mg/day) at week 4, and four tablets (2000 mg/day) at week 6. Doses were decreased, if needed, due to side effects.

ELIGIBILITY:
Inclusion Criteria:

* Men and women ages 18-70 years
* History of mania or hypomania (bipolar I,II, not otherwise specified (NOS) or cyclothymic disorder or schizoaffective disorder/bipolar type)
* Early recovery for cocaine abuse/dependence (between 7 days and 12 weeks of enrollment).
* Any current mood state as indicated by structured diagnostic interview
* No psychotropic medication changes within 7 days prior to enrollment.
* English or Spanish speaking

Exclusion Criteria:

* Pregnant/nursing woman
* Current or past citicoline therapy
* Active suicidal or homicidal ideation with plan and intent
* Dementia, mental retardation or other severe cognitive impairment
* Severe or life threatening medical condition

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2010-07; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: E. Sherwood Brown, PH.D., M.D., Principal Investigator — The UT Southwestern Medical Center of Dallas
Locations (1):
- The UT Southwestern Medical Center of Dallas, Dallas, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from local community behavioral healthcare clinics and through advertising in local publications. The recruitment period was from 5/1/2004 to 4/12/2005.
Pre-assignment Details: Participants were randomized to medication assignment after meeting the inclusion and exclusion criteria and completing the Institutional Review Board(IRB)-approved informed consent process.
Period: Overall Study
Arm/Group | Citicoline | Placebo
Started | 16 (23 completed baseline assessment but 16 completed at least one treatment visit.) | 18 (21 completed baseline assessment but 18 completed at least one treatment visit.)
Completed | 9 (9 completed 12 week trial.) | 4 (4 completed 12 week trial.)
Not Completed | 7 | 14

BASELINE CHARACTERISTICS:
Population: Number of paticipants who completed baseline assessment
Groups:
- Total: Total of all reporting groups
Arm/Group | Citicoline | Placebo | Total
Number analyzed (Participants) | 23 | 21 | 44
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 23 | 21 | 44
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.1 (6.6) | 40.7 (8.0) | 41.4 (7.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 11 | 21
  Male | 13 | 10 | 23
Region of Enrollment [Number; unit: participants]
  United States | 23 | 21 | 44
Inventory of Depressive Symptomatology [Mean (Standard Deviation); unit: Units on a scale] — The IDS-SR is a 30 item self report used to assess the severity of depressive symptoms. The each item has a 4-likert scale, 0 to 3, with 3 representing the worst symptom. The total score of IDS-SR is calculated as a sum of each item score. The range of possible score is between 0 and 90, 0 as no symptom and 90 the worst symptom. The higher the score, the more severe the depression.
  Units on a scale | 43.6 (10.6) | 38.7 (13) | 41.26 (11.9)
Young Mania Rating Scale [Mean (Standard Deviation); unit: Units on a scale] — The YMRS questionnaire has 11 items with scale range 0 to 4 for 7 items and 0 to 8 for 4 items. 0=normal and and 4 or 8 =most abnormal. The total possible score is 0 to 60, 0 being no symptom and 60 the worst symptom. The higher the score, the worse the mania symptoms are.
  Units on a scale | 11.2 (4.9) | 11.5 (7.0) | 11.34 (5.89)
Rey Auditory Verbal Learning Scale [Mean (Standard Deviation); unit: T scores] — The RAVLT consists of 15 nouns read aloud for five consecutive trials with each trial followed by a free-recall trial. The total score is the total number of words recalled through the five trials. Normative RAVLT T-scores was used. the higher T score, the better memory.
  T scores | 36.6 (10.0) | 36.0 (9.0) | 36.33 (9.47)
cocaine used [Number; unit: participants] — Urine drug screen is conducted and if no cocaine is detected in urine, then no cocaine was used. if a positive amount of cocaine is detected in urine, then cocaine was used.
  participants
    No cocaine used | 19 | 19 | 38
    Cocaine used | 4 | 1 | 5
    Unknown | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Cocaine Use Determined by Urine Analysis
Description: Urine drug screens were administered at each visit to detect cocaine in urine. If negative according to urine analysis, it is determined as no cocaine use and if positive, cocaine use. Percentage of participants with no cocaine detected in urine at exit is an outcome measuring treatment effectiveness. Exit week is defined as the last week of treatment. It varied between 2 week an 12 weeks with an average exit week of 10 week and 7 week for the citicoline treatment and placebo groups, respectively. Allowing unequal week of treatment period in measuring outcome enables us to include most participants due to a low retention rate in the end of the study period, 12 weeks.
Time Frame: Biweekly (visit) urine drug screens
Population: Number of participants are those who completed baseline assessment and at least one treatment visit followed by baseline.
Measure: Number; unit: percentage of participants no cocaine
Arm/Group | Citicoline | Placebo
Number analyzed (Participants) | 16 | 18
percentage of participants no cocaine | 62.50 | 50.00
Statistical Analysis 1: Comparison: Citicoline vs Placebo; Null hypothsis is no group association in cocaine use; Test type: Superiority or Other; p = .4637, Chi-squared; df=1 n=34

2. Secondary Outcome: Inventory of Depressive Symptomatology Self Report (IDS-SR).
Description: The IDS-SR is a 30 item self report used to assess the severity of depressive symptoms. The each item has a 4-likert scale, 0 to 3, with 3 representing the worst symptom. The total score of IDS-SR is calculated as a sum of each item score. The range of possible score is between 0 and 90, 0 as no symptom and 90 the worst symptom. The higher the score, the more severe the depression. Exit week is defined as the last week of treatment. It varied between 2 week an 12 weeks with an average exit week of 10 week and 7 week for the citicoline treatment and placebo groups, respectively. Allowing unequal week of treatment period in measuring outcome enables us to include most participants due to a low retention rate in the end of the tudy period, 12 weeks. The outcome was measured by change in scores between baseline and exit (exit - baseline).
Time Frame: Change in scores between baseline and exit (exit - baseline).
Population: Number of participants reported are those who completed baseline assessment and at least one treatment visit.
Measure: Mean (Standard Deviation); unit: units on scale
Arm/Group | Citicoline | Placebo
Number analyzed (Participants) | 16 | 18
units on scale | -20.54 (14.56) | -11.89 (14.45)

3. Secondary Outcome: Young Mania Rating Scale(YMRS).
Description: The YMRS questionnaire has 11 items with scale range 0 to 4 for 7 items and 0 to 8 for 4 items. 0=normal and and 4 or 8 =most abnormal. The total possible score is 0 to 60, 0 being no symptom and 60 the worst symptom. The higher the score, the worse the mania symptoms are. Exit week is defined as the last week of treatment. It varied between 2 week an 12 weeks with an average exit week of 10 week and 7 week for the citicoline treatment and placebo groups, respectively. Allowing unequal week of treatment period in measuring outcome enables us to include most participants due to a low retention rate in the end of the study period, 12 weeks. The outcome was measured by change in scores between baseline and exit (exit - baseline).
Time Frame: Baseline to exit (exit score - baseline score)
Population: Numbers of participants are those who completed baseline assessment and at least one treatment visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Citicoline | Placebo
Number analyzed (Participants) | 16 | 18
units on a scale | -2.00 (8.03) | -2.88 (5.68)

4. Secondary Outcome: Rey Auditory Verbal Learning Test(RAVLT)
Description: The RAVLT consists of 15 nouns read aloud for five consecutive trials with each trial followed by a free-recall trial. The total score is the total number of words recalled through the five trials. Normative RAVLT T-scores was used. the higher T score, the better memory. Exit week is defined as the last week of treatment. It varied between 2 week an 12 weeks with an average exit week of 10 week and 7 week for the citicoline treatment and placebo groups, respectively. Allowing unequal week of treatment period in measuring outcome enables us to include most participants due to a low retention rate in the end of the study period, 12 weeks. The outcome was measured by change in RAVLT T scores between baseline and exit (exit - baseline).
Time Frame: Change in T scores between baseline and exit (exitT score - baseline T score).
Population: number of participants are calculated based on those who completed baseline and at least one treatment visit.
Measure: Mean (Standard Deviation); unit: T score
Arm/Group | Citicoline | Placebo
Number analyzed (Participants) | 16 | 17
T score | 7.06 (11.79) | 3.14 (7.07)

ADVERSE EVENTS:
Arm/Group | Citicoline | Placebo
Serious Adverse Events (participants affected / at risk) | 1/23 | 2/21
Other Adverse Events (participants affected / at risk) | 0/23 | 0/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Citicoline (N=23) | Placebo (N=21)
Skin rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) — The patient discontinued study medication and was scheduled for an exit study visit one week from the event report. Pt. was discontinued from the study.
Hypomania (Psychiatric disorders) | 0 (0) | 1 (1) — Anxiety, paranoia and increased activity and body movements.

LIMITATIONS AND CAVEATS:
Low retention rate in the end of study (12 weeks) leading to a potential underestimation of treatment effectiveness.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No